CLINICAL TRIAL: NCT00489801
Title: RCT Comparing Home-based Cardiac Rehabilitation With Comprehensive Centre-based Cardiac Rehabilitation and Usual Care in Patients Older Than 65 Years With Coronary Heart Disease. The HOMEBASE Trial.
Brief Title: Trial Comparing Home-based Cardiac Rehabilitation With Comprehensive Centre-based Cardiac Rehabilitation in Patients Older Than 65 Years With Coronary Heart Disease. The HOMEBASE Trial
Acronym: HOME-BASE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Velux Fonden (Other)
Responsible Party: Bispebjerg University Hospital, Bispebjerg University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KF 11 2006-4305
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Coronary Heart Disease
Keywords: Cardiac Rehabilitation; Exercise; Heart failure; Coronary heart disease
MeSH Terms: conditions — Coronary Disease; Motor Activity; Heart Failure | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise intervention (Other): Exercise intervention and lifestyle counseling at centre or exercise intervention at home
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise intervention and lifestyle counseling at centre or exercise intervention at home

SUMMARY:
Hypothesis: Home-based cardiac rehabilitation is as effective as comprehensive centre-based cardiac rehabilitation in patients older than 65 years.

DETAILED DESCRIPTION:
Participation in cardiac rehabilitation is known to reduce mortality and morbidity and increase health related quality of life. However, participation rate are low among elderly cardiac patients with coronary heart disease. Home-based cardiac rehabilitation could be an attractive alternative to the centre-based programmes but studies investigating the effect of these programmes are limited and even less is known about the effect among the elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Event of coronary heart disease (new myocardial infarction, CABG or PCI)

Exclusion Criteria:

1. Care home patients.
2. Serious disability incompatible with rehabilitation.
3. Social circumstances incompatible with participation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 115 (Actual)
Dates: Start 2007-01; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | At baseline and after 3,6 and 12 months

SECONDARY OUTCOMES:
Blood pressure, cholesterol, body composition, HRQL | At baseline and after 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bodil Oerkild, MD, ph.d fellow, Principal Investigator
Locations (1):
- Bispebjeg Hospital, Copenhagen, Denmark